CLINICAL TRIAL: NCT03687814
Title: Low FODMAP Plus PEG 3350 for the Treatment of Patients with Irritable Bowel Syndrome-Constipation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Stacy Menees, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00139784
Record Dates: First submitted 2018-09-25; First posted 2018-09-27 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Irritable Bowel Syndrome Characterized by Constipation
MeSH Terms: interventions — FODMAP Diet

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low FODMAP diet plus PEG 3350 (Experimental): Subjects will follow a low FODMAP diet and will take PEG 3350 (Miralax).
  Interventions: Other: Low FODMAP diet/PEG 3350
- Sham diet plus PEG 3350 (Sham Comparator): Subjects will follow a sham diet and will take PEG 3350 (Miralax).
  Interventions: Other: sham diet/PEG 3350

INTERVENTIONS:
Other: Low FODMAP diet/PEG 3350 — Subjects will follow a low FODMAP diet and will take PEG 3350 (Miralax) at 17.7 g (single dose) daily for 4 weeks.
  Other Names: low FODMAP diet
  Arms: Low FODMAP diet plus PEG 3350
Other: sham diet/PEG 3350 — Subjects will follow a sham diet and will take PEG 3350 (Miralax) at 17.7 g (single dose) daily for 4 weeks.
  Other Names: sham diet
  Arms: Sham diet plus PEG 3350

SUMMARY:
Consecutive patients with Irritable Bowel Syndrome with Constipation (IBS-C) will be recruited from the outpatient clinics of the University of Michigan Health System. Eligible patients will be asked to participate in a study that will test the efficacy the PEG 3350 + a diet low in fermentable oligo, di, monosaccharides, and polyols (FODMAP) vs. PEG 3350 plus sham diet. Blinding dietary advice trials is challenging and therefore the sham diet was based on the criteria set forth by Staudacher et al. which emphasizes that the diet must give the impression that is the true intervention diet with similar restrictions, modifications, and time intensity without impacting the intake of essential nutrients, fiber, and FODMAPs. An example of the sham diet's carbohydrates includes: apples, bananas, and pears, and wheat. Oranges, raspberries, strawberries and rice would not be allowed. Additionally, the physicians analyzing the data will be blinded as to which group the patients were randomized.

DETAILED DESCRIPTION:
A. Specific Aims: While a diet low in fermentable oligo, di, monosaccharides and polyols (FODMAPs) has gained popularity as a treatment for patients with Irritable Bowel Syndrome and diarrhea (IBS-D), the impact of this diet on patients with IBS and constipation (IBS-C) is unknown. We propose a randomized, controlled trial in IBS-C patients to compare the efficacy of PEG 3350 and the low FODMAP diet to PEG 3350 and a sham diet. We hypothesize that:

1. The PEG 3350 and low FODMAP diet group will achieve greater improvements in abdominal symptoms including pain, discomfort, and bloating than the group receiving PEG 3350 and the sham diet.
2. The PEG 3350 and low FODMAP diet group will achieve greater improvements in IBS related quality of life and anxiety than the group receiving PEG 3350 and the sham diet.
3. Both strategies will improve constipation related complaints including stool frequency, stool consistency and straining to a similar degree.

We plan to test our central hypothesis and, thereby, accomplish the objective of this application by pursuing the following 2 specific aims:

Aim 1: Compare the proportion of patients with IBS-C on a diet of low FODMAP diet plus PEG 3350 vs. sham diet plus PEG 3350 reporting an improvement of abdominal pain. Our working hypothesis is that a higher proportion of patients randomized to the low FODMAP diet plus PEG 3350 will experience a reduction in the abdominal pain when compared to PEG 3350 plus sham diet alone.

Aim 2: Compare the efficacy of the low FODMAP diet plus PEG 3350 vs. sham diet plus PEG 3350 on pre-specified key clinical and disease specific quality of life endpoints in patients with IBS-C. Through our randomized controlled trial, we will assess the impact of the dietary interventions on stool consistency, stool frequency, and bloating and quality of life endpoints.

A positive result to this study would have significant impact on the treatment of patients with IBS by expanding the indications for the low FODMAP diet to all affected patients, regardless of bowel subtype. This would be particularly relevant to IBS-C patients for whom we currently have few evidence-based diet recommendations outside of increasing fiber intake.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18 and older meeting the Rome IV criteria for IBS-C*:

• Recurrent abdominal pain, on average, at least 1 day/week in the last 3 months, associated with two or more of the following:

1. related to defecation
2. associated with a change in the frequency of stool (reduction of stools)
3. associated with a change in the form of stool (hard or lumpy stools) AND >25% hard stools and <25% loose stools * Criteria fulfilled for the last 3 months

Exclusion Criteria:

* any other IBS subtype other than IBS-C
* >3 spontaneous bowel movements during the last 7 days of run-in
* Have cognitive dysfunction or unable to understand or provide written informed consent
* Pregnancy (evaluated by self-report)
* Comorbid medical problems that may affect gastrointestinal transit or motility:
* Inflammatory bowel disease
* Extra-intestinal disease known to affect the gastrointestinal system (i.e., scleroderma, unstable thyroid disease, etc.)
* Severe renal or hepatic disease
* Previous abdominal surgery other than appendectomy, cholecystectomy, and gynecologic/urologic surgery if performed more than six months prior to enrollment
* Previous treatment with the low FODMAP diet under a dietician guidance
* Concurrent medications not permitted including probiotics, antibiotics, prescription or over-the-counter medication for IBS, and narcotics
* New antidepressant use (less than 3 months on stable dose)
* Active participation in another form of dietary therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2018-11-08 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of abdominal pain as measured by 11-point numerical rating scale | during weeks 3 and 4
  Compare the proportion of patients with IBS-C on a diet of low FODMAP diet plus PEG 3350 vs. sham diet plus PEG 3350 reporting an improvement of abdominal pain. It is defined 30% reduction in abdominal pain during weeks 3 & 4 of each diet compared with baseline using an 11-point numerical rating scale (NRS) (0-no pain, 11-intolerable pain). Appropriate between-group statistical comparisons will be conducted.

SECONDARY OUTCOMES:
Bloating | each treatment week (4 weeks)
  The change in mean score from baseline on the daily 11-point NRS averaged over each treatment week for bloating severity will be compared between the 2 groups.
abdominal discomfort | during weeks 3 and 4
  30% reduction in abdominal discomfort during weeks 3 & 4 of each diet compared with baseline using an 11-point NRS. Appropriate between-group statistical comparisons will be conducted.
Mean number of SBMs per day | week 4
  These will be measured in the last treatment week (the 7-day period before visit 4): The proportion of responders between the 2 groups will be compared. An SBM was defined as a bowel movement that occurred without the use of rescue medication or ≥24 h after the use of rescue medication.
Mean weekly number of spontaneous complete bowel movements | last treatment week
  These will be tallied in the last treatment week (the 7-day period before visit 4):(SCBMs; derived from the number of SBMs without a feeling of incomplete evacuation)
Composite endpoint: Full responder was defined as a patient with >3 SBM per week, an increase of ≥1 SBM per week and >30% pain reduction. | during weeks 3 & 4
  during weeks 3 & 4
stool consistency | Over the 4 weeks of treatment
  a responder will be defined as one who reports an increase in mean daily BSFS value of 1 or more compared to baseline for ≥2 of 4 treatment weeks. The proportion of responders between the 2 groups will be compared. Between group differences in the proportion of patients with an increase in BSFS value of ≥1
Straining | 4 weeks
  The change from baseline in daily numerical rating scale scored as 0 (none), 1 (slight), 2 (mild), 3 (moderate) and 4 (severe) scores averaged over each treatment week for straining will be compared between the 2 groups
IBS-QOL | baseline and week 4
  assess change in IBS-QOL from baseline and the last week of treatment week 4
HADS score | baseline and week 4
  assess change in HADS score from baseline and the last week of treatment of week 4
WPAI questionnaire | baseline and week 4
  assess change in WPAI questionnaire from baseline and the last week of treatment of week 4
Sleep Assessment questionnaire | baseline and week 4
  assess change in Sleep Assessment questionnaire from baseline and the last week of treatment of week 4

CONTACTS AND LOCATIONS:
Overall Officials: Stacy B Menees, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States